CLINICAL TRIAL: NCT01815255
Title: Efficacy and Safety Evaluation of TDF-based Regimen in Thai HIV-infected Children
Brief Title: TDF Long Term Study
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Bamrasnaradura Infectious Diseases Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 133
Record Dates: First submitted 2013-02-07; First posted 2013-03-21 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV-infected Thai Children
Keywords: TDF-based regimen; HIV-infected children; Thai; generic; safety and efficacy; renal status; To assess effect of TDF on renal problem in HIV-infected children receiving TDF-based once daily regimen; To compare the effectiveness and clinical usefulness of different tools of adherence
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Phlebotomy will be for safety evaluation and will be drawn according to the schedule of visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tenofovir (TDF): HIV-infected children who are currently on TDF-based regimen or are changing to TDF based on their clinical indication
  Interventions: Drug: tenofovir (TDF)

INTERVENTIONS:
Drug: tenofovir (TDF)

SUMMARY:
This study will assess the safety and efficacy of generic TDF from Governmental Pharmaceutical Organization (GPO) in HIV-infected children

DETAILED DESCRIPTION:
TDF is a nucleotide reverse transcriptase inhibitor (NRTI) which can be taken only once per day and continues to have good efficacy even in patients who have resistance to other NNRTI in the absence of K65R mutation. TDF is a choice for patients with NRTI resistance, or those that require once-daily regimen to improve adherence. Currently, TDF has not been approved by the US FDA for children less than 18 years, but pediatricians has been using TDF in children who have treatment failure because of limitation of a more appropriate pediatric ARV. The Thai national guideline for pediatric 2009 recommend the use of TDF in children who have failed the first line therapy with multi-NRTI mutation and are more than 30 kilograms or have tanner stage 4 or more. However, the problem is that there is no pediatric TDF formulation. The available preparation of 300 mg tear drop tablet, if cut in half, may increase dosing errors, more or less by 18-37%. This will affect the blood level and/or toxicities. Therefore, the Thai Governmental Pharmaceutical Organization (GPO) has produced a generic TDF formulation that can be used in HIV-infected children. This study will assess the safety and efficacy information in children using this generic pediatric TDF formulation.

ELIGIBILITY:
Inclusion Criteria:

* children who are changing to TDF due to adherence problem or treatment failure
* children who are already on TDF due to their clinical indication

Exclusion Criteria:

* child/caretaker refuse to participate in this study
* cannot adhere to the study schedule

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-infected children who are currently taking or are changing to tenofovir-(TDF) based regimen
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
viral load | week 48 and 96
  Number of patients who have viral load less than 50 copies/ml at week 48 and week 96

SECONDARY OUTCOMES:
renal status | weeks 24, 48, 72, and 96
  Number of patients with renal toxicity assessed by GFR and with proximal tubular effect
adherence | every 3 months
  Agreement between self reported adherence by visual analogue scale (VAS) pill count and TDM Sensitivity and specificity of self-reported adherence and pill count against gold standards of TDM and undetectable viral load
resistance | every 3 months
  Resistant mutations in patients who fail TDF-based regimen and response to new regimen
adverse events | weeks 24, 48, 72, and 96
  Proportion of patients who develop adverse events which are related to TDF and other ARVs

CONTACTS AND LOCATIONS:
Overall Officials: Wasana Prasitsuebsai, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration; Jurai Wongsawat, MD, Principal Investigator — Bamrasnadura Institute
Locations (2):
- Thailand (2):
  - HIV-NAT, Bangkok
  - King Chulalongkorn Hospital, Chulalongkorn University, Bangkok

REFERENCES:
- [Result] Prasitsuebsai W, Puthanakit T, Apornpong T, Keadpudsa S, Bunupuradah T, Chuanjaroen T, Thammajaruk N, Jupimai T, Kerr SJ, Ananworanich J. Bone and Renal Safety at 96 weeks of TDF-containing in HIV-infected Thai children. Abstract # 905 presented at the 21st CROI 2014, March 3-6, 2014 at Boston, USA
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)'s website — http://www.hivnat.org